CLINICAL TRIAL: NCT03979313
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of MEDI8897, a Monoclonal Antibody With an Extended Half-life Against Respiratory Syncytial Virus, in Healthy Late Preterm and Term Infants (MELODY)
Brief Title: A Study to Evaluate the Safety and Efficacy of MEDI8897 for the Prevention of Medically Attended Lower Respiratory Tract Infection Due to Respiratory Syncytial Virus in Healthy Late Preterm and Term Infants (MELODY)
Acronym: MELODY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D5290C00004; 2019-000114-11 (EudraCT Number); NCT05238974 (obsolete NCT alias)
Record Dates: First submitted 2019-05-30; First posted 2019-06-07 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus; RSV; Late Preterm Infants; Healthy Infants; Lower Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI8897 (Experimental): Anti-RSV monoclonal antibody with an extended half-life
  Interventions: Drug: MEDI8897
- Placebo (Placebo Comparator): Commercially available 0.9% (w/v) saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI8897 — Anti-RSV monoclonal antibody with an extended half-life
  Arms: MEDI8897
Drug: Placebo — Commercially available 0.9% (w/v) saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, pharmacokinetics (PK), and antidrug antibody (ADA) response for MEDI8897 in healthy late preterm and term infants who are 35 weeks or greater gestational age and entering their first RSV season.

DETAILED DESCRIPTION:
This pivotal Phase 3 study will determine if MEDI8897 will prevent medically attended RSV-confirmed lower respiratory tract infections (LRTI) in healthy infants entering their first RSV season. The population to be enrolled is healthy late preterm and term infants born 35 weeks 0 days or greater gestational age (GA) who would not be eligible to receive RSV prophylaxis. A total of approximately 3,000 infants will be randomized 2:1 to receive either MEDI8897 or placebo. All subjects will be followed for approximately 510 days after dosing. Enrollment is planned at approximately 350 sites across the USA, Canada, Europe, Asia, and Southern Hemisphere.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy infants in their first year of life and born at or after 35 weeks 0 days GA
* Infants who are entering their first RSV season at the time of screening

Key Exclusion Criteria:

* Meets national or other local criteria to receive commercial palivizumab
* Any fever (≥ 100.4°F [≥ 38.0°C], regardless of route) or acute illness within 7 days prior to randomization
* Active RSV infection (a child with signs/symptoms of respiratory infection must have negative RSV testing) or known prior history of RSV infection
* Receipt of palivizumab or other RSV monoclonal antibody or any RSV vaccine, including maternal RSV vaccination

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3012 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (176):
- United States (62):
  - Research Site, Birmingham, Alabama
  - Research Site, Fort Defiance, Arizona
  - Research Site, Fayetteville, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Downey, California
  - Research Site, National City, California
  - Research Site, Paramount, California
  - Research Site, West Covina, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Fort Gordon, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Bardstown, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Jackson, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Gallup, New Mexico
  - Research Site, Shiprock, New Mexico
  - Research Site, Syracuse, New York
  - Research Site, Boone, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Erie, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, North Charleston, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Kingsport, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Baytown, Texas
  - Research Site, Dallas, Texas
  - Research Site, Edinburg, Texas
  - Research Site, League City, Texas
  - Research Site, Longview, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas
  - Research Site, Layton, Utah
  - Research Site, Roy, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, South Jordan, Utah
  - Research Site, St. George, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Marshfield, Wisconsin
- Research Site, San Miguel de Tucumán, Argentina
- Australia (2):
  - Research Site, Clayton
  - Research Site, Nedlands
- Austria (2):
  - Research Site, Graz
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Ghent
- Bulgaria (7):
  - Research Site, Montana
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Pierrefonds, Quebec
- Research Site, Santiago, Chile
- Colombia (5):
  - Research Site, Cali
  - Research Site, Chía
  - Research Site, Medellín
  - Research Site, Montería
  - Research Site, Soledad
- Research Site, Havlíčkův Brod, Czechia
- Estonia (3):
  - Research Site, Paide
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (9):
  - Research Site, Espoo
  - Research Site, Helsinki
  - Research Site, Jarvenpaa
  - Research Site, Kokkola
  - Research Site, Oulu
  - Research Site, Pori
  - Research Site, Seinäjoki
  - Research Site, Tampere
  - Research Site, Turku
- France (7):
  - Research Site, Amiens
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Créteil
  - Research Site, Lille
- Germany (3):
  - Research Site, Frankenthal
  - Research Site, Leipzig
  - Research Site, Mannheim
- Israel (2):
  - Research Site, Beersheba
  - Research Site, Netanya
- Research Site, Roma, Italy
- Japan (8):
  - Research Site, Fukuyama-shi
  - Research Site, Kawasaki-shi
  - Research Site, Maebashi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Shizuoka
  - Research Site, Yokosuka-shi
- Latvia (3):
  - Research Site, Jēkabpils
  - Research Site, Riga
  - Research Site, Valmiera
- Research Site, Kaunas, Lithuania
- Research Site, México, Mexico
- New Zealand (4):
  - Research Site, Christchurch
  - Research Site, Grafton
  - Research Site, Papatoetoe
  - Research Site, Wellington
- Panama (4):
  - Research Site, Cuidad de Panama
  - Research Site, David
  - Research Site, La Chorrera
  - Research Site, Panama City
- Poland (4):
  - Research Site, Krakow
  - Research Site, Torun
  - Research Site, Wroclaw
  - Research Site, Łęczna
- Russia (2):
  - Research Site, Perm
  - Research Site, Saint Petersburg
- South Africa (6):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Pretoria
  - Research Site, Rondebosch
  - Research Site, Soweto
- South Korea (2):
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (16):
  - Research Site, Alicante
  - Research Site, Antequera
  - Research Site, Castellon
  - Research Site, Córdoba
  - Research Site, Granada
  - Research Site, Leganés
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Móstoles
  - Research Site, Pozuelo de Alarcón
  - Research Site, San Cristóbal de La Laguna
  - Research Site, Sant Cugat del Vallès
  - Research Site, Sant Joan d'Alacant
  - Research Site, Santiago de Compostela
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Linköping
  - Research Site, Stockholm
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Izmir
  - Research Site, Kocaeli
- Ukraine (5):
  - Research Site, Chernivtsі
  - Research Site, Dnipro
  - Research Site, Kyiv
  - Research Site, Sumy
  - Research Site, Vinnytsia
- United Kingdom (2):
  - Research Site, Liverpool
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bolanos R, Araos R, Gonzalez C, Sepulveda D, Falconi JF, Averin A, Atwood M, Quinn E, Law AW, Mendes D. Cost-effectiveness of strategies using preventive interventions to protect infants in Chile from respiratory syncytial virus. Expert Rev Vaccines. 2025 Dec;24(1):904-913. doi: 10.1080/14760584.2025.2562201. Epub 2025 Oct 2. PMID 40958705
- [Derived] Arbetter D, Gopalakrishnan V, Aksyuk AA, Ahani B, Chang Y, Dagan R, Esser MT, Hammitt LL, Mankad VS, Saez-Llorens X, Shen D, Leach A, Kelly EJ, Villafana T, Wilkins D. Lower Respiratory Tract Infections Following Respiratory Syncytial Virus Monoclonal Antibody Nirsevimab Immunization Versus Placebo: Analysis From a Phase 3 Randomized Clinical Trial (MELODY). Clin Infect Dis. 2025 Oct 6;81(3):634-644. doi: 10.1093/cid/ciae596. PMID 39656748
- [Derived] Langer S, Holzapfel S, August L, Badura A, Wellmann S, Mack I. Parental knowledge and attitudes to infant immunization in the context of RSV: All about confidence? Vaccine. 2024 Oct 3;42(23):126050. doi: 10.1016/j.vaccine.2024.06.018. Epub 2024 Jun 19. PMID 38902186
- [Derived] Dagan R, Hammitt LL, Seoane Nunez B, Baca Cots M, Bosheva M, Madhi SA, Muller WJ, Zar HJ, Chang Y, Currie A, Grenham A, Shroff M, Takas T, Mankad VS, Leach A, Villafana T. Infants Receiving a Single Dose of Nirsevimab to Prevent RSV Do Not Have Evidence of Enhanced Disease in Their Second RSV Season. J Pediatric Infect Dis Soc. 2024 Feb 26;13(2):144-147. doi: 10.1093/jpids/piad113. PMID 38219024
- [Derived] Ahani B, Tuffy KM, Aksyuk AA, Wilkins D, Abram ME, Dagan R, Domachowske JB, Guest JD, Ji H, Kushnir A, Leach A, Madhi SA, Mankad VS, Simoes EAF, Sparklin B, Speer SD, Stanley AM, Tabor DE, Hamren UW, Kelly EJ, Villafana T. Molecular and phenotypic characteristics of RSV infections in infants during two nirsevimab randomized clinical trials. Nat Commun. 2023 Jul 19;14(1):4347. doi: 10.1038/s41467-023-40057-8. PMID 37468530
- [Derived] Muller WJ, Madhi SA, Seoane Nunez B, Baca Cots M, Bosheva M, Dagan R, Hammitt LL, Llapur CJ, Novoa JM, Saez Llorens X, Grenham A, Kelly EJ, Mankad VS, Shroff M, Takas T, Leach A, Villafana T; MELODY Study Group. Nirsevimab for Prevention of RSV in Term and Late-Preterm Infants. N Engl J Med. 2023 Apr 20;388(16):1533-1534. doi: 10.1056/NEJMc2214773. Epub 2023 Apr 5. No abstract available. PMID 37018470
- [Derived] Hammitt LL, Dagan R, Yuan Y, Baca Cots M, Bosheva M, Madhi SA, Muller WJ, Zar HJ, Brooks D, Grenham A, Wahlby Hamren U, Mankad VS, Ren P, Takas T, Abram ME, Leach A, Griffin MP, Villafana T; MELODY Study Group. Nirsevimab for Prevention of RSV in Healthy Late-Preterm and Term Infants. N Engl J Med. 2022 Mar 3;386(9):837-846. doi: 10.1056/NEJMoa2110275. PMID 35235726
- [Derived] Ginsburg AS, Srikantiah P. Respiratory syncytial virus: promising progress against a leading cause of pneumonia. Lancet Glob Health. 2021 Dec;9(12):e1644-e1645. doi: 10.1016/S2214-109X(21)00455-1. Epub 2021 Nov 11. No abstract available. PMID 34774184
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00004&attachmentIdentifier=2d401e07-a37e-411e-8084-97fddbc8a78e&fileName=D5290C00004_-_Protocol_Redacted_9aug2023_a.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00004&attachmentIdentifier=8b9437c7-c329-4235-8ace-9247ca221eed&fileName=D5290C00004_-_Statistical_Analysis_Plan_Redacted_9aug2023_a.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00004&attachmentIdentifier=d2412c63-3b47-4c1e-a808-4f171d42b52a&fileName=d5290c00004-study-synopsis-Redacted-9aug2023_a.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject In: 23-07-2019. Last Subject Last Visit: 21-03-2023. The study was planned to analyze data on the full enrolment of approximately 3000 infants. The impact of the COVID-19 pandemic on RSV circulation led to the decision to analyze the primary endpoint based on the first 1500 subjects enrolled (Primary Cohort). After the COVID-19 pandemic the study restarted. So the study comprised 2 cohorts: a Primary and a Safety for a total of 3319 screened subjects.
Pre-assignment Details: 1626 screened subjects in Primary Cohort. 136 subjects did not start the study: 98 not meeting the I/E criteria, 6 lost to follow-up, 25 withdrew the informed consent, 7 for other reason.
  Overall 3319 screened subjects. 307 did not start the study: 192 not meeting the I/E criteria, 11 lost to follow-up, 90 withdrew the informed consent, 14 for other reason.
Groups:
- Placebo; Medi8897: Single IM dose of 50 mg (if < 5 kg weight at time of dosing) or 100 mg (if ≥ 5 kg weight at time of dosing).
Period: Primary Cohort (Data Cut Off 11/3/2021)
Arm/Group | Placebo | Medi8897
Started | 496 | 994
Completed Day 151 Follow up | 488 | 977
Completed Day 361 Follow up | 453 | 914
Treated Participants | 491 | 994
Completed (Study completion at Day 511. At this DCO several subjects did not complete the study and were still ongoing.) | 43 | 89
Not Completed | 453 | 905
Not completed — Lost to Follow-up | 3 | 9
Not completed — Any Other Reason | 3 | 4
Not completed — Death | 0 | 4
Not completed — Withdrawal by Subject | 14 | 20
Not completed — Covid-19 pandemic | 1 | 3
Not completed — Ongoing at the DCO date | 432 | 865
Period: All Subjects
Arm/Group | Placebo | Medi8897
Started | 1003 | 2009
Completed Day 151 Follow up | 985 | 1977
Completed Day 361 Follow up | 967 | 1944
Treated Participants | 997 | 1997
Completed (Study completion at day 511) | 923 | 1873
Not Completed | 80 | 136
Not completed — Any Other Reason | 16 | 23
Not completed — Covid-19 | 1 | 3
Not completed — Withdrawal by Subject | 35 | 44
Not completed — Death | 0 | 5
Not completed — Lost to Follow-up | 28 | 61

BASELINE CHARACTERISTICS:
Population: These are the Overall Number of All Subjects Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Medi8897 | Total
Number analyzed (Participants) | 1003 | 2009 | 3012
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Two analysis population data are shown: Primary Cohort and All Subjects
  Months
    Age (months) in Primary Cohort: number analyzed (Participants) | 496 | 994 | 1490
    Age (months) in Primary Cohort | 3.012 (2.2520) | 2.912 (2.2099) | 2.946 (2.2237)
    Age (months) in All Subjects | 2.918 (2.2740) | 2.905 (2.220) | 2.909 (2.2376)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two analysis population data are shown: Primary Cohort and All Subjects
  Participants
    Sex in Primary Cohort: number analyzed (Participants) | 496 | 994 | 1490
    Sex in Primary Cohort: Female | 257 | 464 | 721
    Sex in Primary Cohort: Male | 239 | 530 | 769
    Sex in All Subjects: Female | 500 | 938 | 1438
    Sex in All Subjects: Male | 503 | 1071 | 1574
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Two analysis population data are shown; Primary Cohort and All Subjects 3 subjects in the Medi998 had missing value for Race
  Participants
    Race in Primary Cohort: number analyzed (Participants) | 496 | 994 | 1490
    Race in Primary Cohort: American Indian or Alaska Native | 26 | 57 | 83
    Race in Primary Cohort: Asian | 18 | 36 | 54
    Race in Primary Cohort: Black or African American | 136 | 286 | 422
    Race in Primary Cohort: Native Hawaiian or other Pacific Islander | 5 | 6 | 11
    Race in Primary Cohort: White | 272 | 524 | 796
    Race in Primary Cohort: Multiple categories checked | 1 | 12 | 13
    Race in Primary Cohort: Other | 38 | 70 | 108
    Race in Primary Cohort: Missing | 0 | 3 | 3
    Race in All Subjects: American Indian or Alaska Native | 52 | 92 | 144
    Race in All Subjects: Asian | 50 | 109 | 159
    Race in All Subjects: Black or African American | 138 | 299 | 437
    Race in All Subjects: Native Hawaiian or other Pacific Islander | 8 | 15 | 23
    Race in All Subjects: White | 541 | 1052 | 1593
    Race in All Subjects: Multiple categories checked | 8 | 19 | 27
    Race in All Subjects: Other | 206 | 420 | 626
    Race in All Subjects: Missing | 0 | 3 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With MA RSV LRTI With Hospitalisation Through 150 Days Post Dose (Primary Cohort)
Description: Hospitalization Analysed on Primary Cohort Through 150 Days (N=1490 Participants)
Time Frame: Through 150 Days Post Dose
Population: ITT population / Primary Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Medi8897
Number analyzed (Participants) | 496 | 994
Participants
  Observed events through day 150 post dose | 8 | 6
  Subjects requiring imputation (subjects without events and not followed through 150 days post dose) | 6 | 15
  Subjects without event through day 150 post dose | 482 | 973
Statistical Analysis 1: Comparison: Placebo vs Medi8897; Test type: Superiority; p = 0.0708, Poisson Model; Relative Risk Reduction (RRR) = 62.15, 95% CI 2-sided [-8.57 to 86.80] — RRR of Medi8897 versus placebo; 95% CI and p-value estimated with Poisson regression with robust variance (including stratification factors [age at randomisation] as covariate) obtained after multiple imputation

2. Primary Outcome: Number of Participants With MA RSV LRTI Through 150 Days Post Dose (Primary Cohort)
Description: Primary Endpoint Analysed on Primary Cohort Through 150 Days (N=1490 Participants)
Time Frame: Through 150 Days Post Dose
Population: ITT population / Primary Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Medi8897
Number analyzed (Participants) | 496 | 994
Participants
  Observed events through day 150 post dose | 25 | 12
  Subjects requiring imputation (Subjects without events and not followed through 150 days post dose) | 6 | 15
  Subjects without event through day 150 post dose | 465 | 967
Statistical Analysis 1: Comparison: Placebo vs Medi8897; Test type: Superiority; p < 0.0001, Poisson Model; Relative Risk Reduction (RRR) = 74.53, 95% CI 2-sided [49.63 to 87.12] — [estimate comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Number of Participants With MA RSV LRTI Through 150 Days Post Dose (All Subjects)
Description: Primary Endpoint Analysed on All Subjects Through 150 Days (N=3012 participants)
Time Frame: Through 150 Days Post Dose
Population: ITT population / All Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Medi8897
Number analyzed (Participants) | 1003 | 2009
Participants
  Observed events through day 150 post dose | 54 | 24
  Subjects requiring imputation (Subjects without events and not followed through 150 days post dose) | 17 | 31
  Subjects without event through day 150 post dose | 932 | 1954
Statistical Analysis 1: Comparison: Placebo vs Medi8897; Test type: Superiority; p < 0.0001, Poisson Model; Relative Risk Reduction (RRR) = 76.36, 95% CI 2-sided [62.27 to 85.18] — [estimate comment as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Number of Participants With MA RSV LRTI With Hospitalisation Through 150 Days Post Dose (All Subjects)
Description: Hospitalization Analysed on All Subjects Through 150 Days (N=3012 participants)
Time Frame: Through 150 Days Post Dose
Population: ITT population / All Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Medi8897
Number analyzed (Participants) | 1003 | 2009
Participants
  Observed events through day 150 post dose | 20 | 9
  Subjects requiring imputation (Subjects without events and not followed through 150 days post dose) | 18 | 31
  Subjects without event through day 150 post dose | 965 | 1969
Statistical Analysis 1: Comparison: Placebo vs Medi8897; Test type: Superiority; p = 0.0002, Poisson Model; Relative Risk Reduction (RRR) = 76.84, 95% CI 2-sided [49.36 to 89.41] — [estimate comment as in outcome 1, analysis 1]

5. Other Pre Specified Outcome: Number of Participants With Disease From the 2nd RSV Season (All Subjects)
Time Frame: From Day 361 to Day 510 Post Dose
Population: ITT population / All Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Medi8897
Number analyzed (Participants) | 967 | 1944
Participants
  MA RSV LRTI (protocol defined) | 10 | 19
  MA RSV LRTI hospitalisation (protocol defined) | 3 | 3

6. Secondary Outcome: Summary of Serum Concentrations (ug/mL) of MEDI8897 by Group
Description: Number of Subjects with at Least one Assessment
Time Frame: By visit until day 360 post dose
Population: As Treated Population (1997 Participants Treated in MEDI8897 arm)/ All Subjects
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- Medi8897, 50 mg: Subjects with Weight < 5 Kg
- Medi8897, 100 mg: Subjects with Weight >= 5 Kg
Arm/Group | Medi8897, 50 mg | Medi8897, 100 mg
Number analyzed (Participants) | 799 | 1198
ug/mL
  Day 7 Post Dose: number analyzed (Participants) | 40 | 59
  Day 7 Post Dose | 89.91 (39.3) | 164.03 (15.8)
  Day 14 Post Dose: number analyzed (Participants) | 264 | 264
  Day 14 Post Dose | 74.09 (124.9) | 105.05 (89.2)
  Day 30 Post Dose: number analyzed (Participants) | 470 | 878
  Day 30 Post Dose | 68.63 (58.6) | 100.54 (90.1)
  Day 150 Post Dose: number analyzed (Participants) | 618 | 969
  Day 150 Post Dose | 18.32 (63.1) | 27.73 (62.9)
  Day 360 Post Dose: number analyzed (Participants) | 659 | 1001
  Day 360 Post Dose | 1.75 (76.7) | 2.86 (85.7)

7. Secondary Outcome: Anti-drug Antibody Results by Visit (As Treated Population)
Description: Number of subjects with a positive result and a valid titer result at the specific visit
Time Frame: From baseline to 360 day post dose visit
Population: As Treated Population / All Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Medi8897
Number analyzed (Participants) | 968 | 1926
Participants
  Baseline | 4 | 4
  Day 30 Post Dose: number analyzed (Participants) | 705 | 1370
  Day 30 Post Dose | 2 | 14
  Day 150 Post Dose: number analyzed (Participants) | 885 | 1765
  Day 150 Post Dose | 1 | 21
  Day 360 Post Dose: number analyzed (Participants) | 862 | 1778
  Day 360 Post Dose | 10 | 81

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed up to 510 days post dose . Adverse Events monitored/assessed up to day 360 post dose.
Description: Treatment Emergent Adverse Events through 360 days post dose are reported for Placebo and Medi8897 arms. The data are for the Treated Participants (997 for Placebo and 1997 for Medi8897 arm).
Arm/Group | Placebo | MEDI8897
All-Cause Mortality (participants affected / at risk) | 0/997 | 5/1997
Serious Adverse Events (participants affected / at risk) | 83/997 | 149/1997
Other Adverse Events (participants affected / at risk) | 836/997 | 1717/1997
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=997) | MEDI8897 (N=1997)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Fever neonatal (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 6 (6)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Abscess of external auditory meatus (Infections and infestations) | 1 (1) | 0 (0)
Adenoviral upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Botulism (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 17 (18) | 27 (28)
Bronchitis (Infections and infestations) | 4 (5) | 3 (5)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 3 (5)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1)
Bronchogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Exanthema subitum (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5) | 14 (15)
Gastroenteritis escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 3 (3) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 6 (7)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 13 (14)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia viral (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 10 (10) | 5 (5)
Respiratory syncytial virus bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 5 (5) | 7 (7)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4)
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Phenylketonuria (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Dairy intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Food refusal (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 4 (4)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Idiopathic generalised epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Behavioural insomnia of childhood (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep terror (Psychiatric disorders) | 0 (0) | 1 (1)
Staring (Psychiatric disorders) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Kawasaki's disease (Vascular disorders) | 1 (1) | 2 (2)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Allergic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Allergic gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=997) | MEDI8897 (N=1997)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Faeces soft (Gastrointestinal disorders) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 4 (4) | 13 (13)
Food protein-induced enterocolitis syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 (14) | 31 (32)
Gingival cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (3) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 5 (6) | 2 (2)
Infant dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 11 (13) | 41 (41)
Infantile spitting up (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 7 (7)
Teething (Gastrointestinal disorders) | 70 (85) | 138 (171)
Toothache (Gastrointestinal disorders) | 1 (1) | 6 (12)
Umbilical hernia (Gastrointestinal disorders) | 4 (4) | 14 (14)
Vomiting (Gastrointestinal disorders) | 32 (35) | 59 (63)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Crying (General disorders) | 0 (0) | 1 (1)
Developmental delay (General disorders) | 0 (0) | 3 (3)
Discomfort (General disorders) | 2 (2) | 10 (10)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 4 (4) | 2 (2)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 4 (4)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
Mass (General disorders) | 0 (0) | 2 (2)
Pfapa syndrome (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 122 (165) | 290 (378)
Secretion discharge (General disorders) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 2 (2)
Vaccination site pain (General disorders) | 1 (1) | 3 (5)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1)
Vaccination site swelling (General disorders) | 0 (0) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Xerosis (General disorders) | 1 (1) | 5 (6)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 7 (7)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 6 (6)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 9 (9)
Dust allergy (Immune system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 18 (22) | 30 (36)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Milk allergy (Immune system disorders) | 4 (7) | 7 (7)
Multiple allergies (Immune system disorders) | 1 (1) | 2 (2)
Reaction to preservatives (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 6 (6) | 8 (8)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 2 (2) | 2 (2)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 3 (3) | 2 (2)
Abscess neck (Infections and infestations) | 1 (1) | 1 (1)
Acarodermatitis (Infections and infestations) | 15 (20) | 32 (39)
Acute sinusitis (Infections and infestations) | 3 (3) | 2 (2)
Adenoviral upper respiratory infection (Infections and infestations) | 0 (0) | 6 (6)
Adenovirus infection (Infections and infestations) | 3 (3) | 1 (1)
Amoebiasis (Infections and infestations) | 0 (0) | 3 (3)
Aorta hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Amoebic dysentery (Infections and infestations) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Ascariasis (Infections and infestations) | 0 (0) | 1 (1)
Asymptomatic covid-19 (Infections and infestations) | 7 (8) | 8 (8)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 12 (14) | 20 (22)
Borrelia infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 71 (86) | 119 (139)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 31 (34) | 60 (76)
Bronchitis viral (Infections and infestations) | 2 (3) | 1 (1)
Bullous impetigo (Infections and infestations) | 1 (1) | 5 (5)
Covid-19 (Infections and infestations) | 59 (62) | 97 (98)
Candida infection (Infections and infestations) | 5 (5) | 4 (5)
Candida nappy rash (Infections and infestations) | 3 (3) | 19 (19)
Cellulitis (Infections and infestations) | 3 (3) | 6 (6)
Citrobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 56 (61) | 137 (157)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 13 (13)
Brachycephaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 2 (3) | 6 (6)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 3 (3)
Croup infectious (Infections and infestations) | 7 (7) | 17 (18)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Dacryocanaliculitis (Infections and infestations) | 0 (0) | 2 (2)
Dacryocystitis (Infections and infestations) | 3 (3) | 2 (2)
Dermatitis infected (Infections and infestations) | 1 (1) | 1 (1)
Dermatophytosis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 2 (2) | 1 (1)
Bronchogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 4 (5) | 4 (4)
Ear infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Ear lobe infection (Infections and infestations) | 1 (1) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 2 (2)
Enterobiasis (Infections and infestations) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 4 (5)
Exanthema subitum (Infections and infestations) | 27 (27) | 30 (30)
Eye infection (Infections and infestations) | 1 (1) | 7 (9)
Buried penis syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 2 (2)
Folliculitis (Infections and infestations) | 4 (4) | 14 (15)
Fungal infection (Infections and infestations) | 1 (1) | 2 (2)
Fungal skin infection (Infections and infestations) | 19 (19) | 35 (37)
Furuncle (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 100 (113) | 202 (246)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Congenital anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastroenteritis enteroviral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 8 (11) | 21 (23)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 1 (2)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 3 (3)
Genital candidiasis (Infections and infestations) | 1 (1) | 2 (2)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Gianotti-crosti syndrome (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 19 (19) | 42 (43)
Congenital nystagmus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Helminthic infection (Infections and infestations) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 3 (3) | 5 (5)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 2 (2) | 5 (5)
Human herpesvirus 6 infection (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 31 (35) | 43 (47)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Congenital tongue anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 9 (10)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 9 (9) | 35 (37)
Lice infestation (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 34 (44) | 47 (69)
Lower respiratory tract infection viral (Infections and infestations) | 12 (12) | 9 (9)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Measles (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Congenital torticollis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 9 (10)
Nasopharyngitis (Infections and infestations) | 237 (471) | 441 (946)
Omphalitis (Infections and infestations) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 22 (23) | 55 (60)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 4 (4)
Oral infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 6 (6) | 6 (6)
Otitis media (Infections and infestations) | 76 (111) | 154 (218)
Congenital vesicoureteric reflux (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 44 (53) | 82 (126)
Otitis media chronic (Infections and infestations) | 1 (2) | 2 (2)
Parasitic gastroenteritis (Infections and infestations) | 2 (2) | 4 (4)
Paronychia (Infections and infestations) | 2 (2) | 11 (12)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 28 (28) | 72 (80)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 9 (9) | 16 (16)
Pneumonia (Infections and infestations) | 6 (6) | 11 (11)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia moraxella (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Pustule (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 1 (1) | 3 (3)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 3 (3) | 16 (16)
Pyoderma streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 2 (2)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 14 (14) | 13 (13)
Respiratory syncytial virus bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 102 (146) | 201 (272)
Rhinolaryngitis (Infections and infestations) | 0 (0) | 1 (1)
Roseola (Infections and infestations) | 14 (14) | 24 (24)
Anaemia neonatal (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 7 (7) | 9 (9)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 2 (2)
Skin candida (Infections and infestations) | 3 (3) | 9 (9)
Skin infection (Infections and infestations) | 2 (3) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 3 (3) | 2 (2)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 4 (4) | 4 (4)
Subglottic laryngitis (Infections and infestations) | 2 (3) | 1 (1)
Suspected covid-19 (Infections and infestations) | 7 (7) | 10 (10)
Tinea capitis (Infections and infestations) | 3 (3) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 4 (4)
Tinea pedis (Infections and infestations) | 1 (1) | 1 (1)
Tinea versicolour (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 7 (7) | 14 (15)
Tracheitis (Infections and infestations) | 2 (2) | 4 (4)
Tracheobronchitis (Infections and infestations) | 3 (3) | 2 (2)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 316 (621) | 639 (1316)
Urinary tract infection (Infections and infestations) | 14 (15) | 22 (26)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Vaccination site infection (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 10 (10) | 22 (22)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 2 (2)
Viral diarrhoea (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 21 (22) | 35 (36)
Viral pharyngitis (Infections and infestations) | 2 (2) | 9 (9)
Klippel-feil syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 30 (32) | 85 (90)
Viral rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Viral tonsillitis (Infections and infestations) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 60 (77) | 132 (162)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 22 (24) | 27 (31)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 4 (4)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Chemical burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 11 (11)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Macrocephaly (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in ear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mitochondrial encephalomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in throat (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foreign body ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gingival injury (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 6 (7) | 16 (17)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Oral contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Radial head dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 8 (8)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 5 (5) | 9 (10)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 3 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 34 (47) | 72 (90)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood copper increased (Investigations) | 0 (0) | 1 (1)
Blood immunoglobulin e increased (Investigations) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 7 (8) | 13 (13)
Plagiocephaly (Congenital, familial and genetic disorders) | 4 (4) | 11 (11)
Blood lead increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 5 (5)
Cardiac murmur (Investigations) | 4 (4) | 5 (5)
Cardiac murmur functional (Investigations) | 0 (0) | 1 (1)
Echocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 2 (2)
Medical observation normal (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Sars-cov-2 test negative (Investigations) | 27 (30) | 48 (58)
Sars-cov-2 test positive (Investigations) | 4 (4) | 3 (3)
Transaminases increased (Investigations) | 0 (0) | 2 (2)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Breast milk substitute intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dairy intolerance (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Poor feeding infant (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Telangiectasia congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Head deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vascular malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rib deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Cartilage neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 9 (9)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Chorea (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 5 (5) | 4 (4)
Gross motor delay (Nervous system disorders) | 1 (1) | 3 (3)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Horner's syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Hypertonia (Nervous system disorders) | 1 (1) | 1 (1)
Hypotonia (Nervous system disorders) | 2 (2) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Idiopathic partial epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Infant irritability (Nervous system disorders) | 4 (4) | 1 (1)
Motor developmental delay (Nervous system disorders) | 0 (0) | 2 (2)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1)
Post-traumatic epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Seizure like phenomena (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Speech disorder developmental (Nervous system disorders) | 0 (0) | 3 (3)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 3 (3)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Irritability (Psychiatric disorders) | 11 (11) | 22 (26)
Poor quality sleep (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 7 (8) | 12 (14)
Sleep disorder (Psychiatric disorders) | 1 (1) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesicoureteric reflux (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Balanoposthitis (Reproductive system and breast disorders) | 2 (2) | 6 (6)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Genital discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital labial adhesions (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Genital pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile adhesion (Reproductive system and breast disorders) | 5 (5) | 6 (6)
Penile discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal adhesion (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 8 (8) | 14 (14)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Brief resolved unexplained event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 13 (13)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Childhood asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 58 (69) | 115 (145)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 86 (113) | 164 (208)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 18 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 13 (14)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 65 (85) | 152 (216)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (8)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (11)
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 12 (15)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Acne infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dandruff (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 21 (22) | 44 (44)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (12)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 25 (28) | 56 (59)
Astigmatism (Eye disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 16 (18) | 39 (41)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 103 (118) | 224 (267)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 19 (19) | 39 (41)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 52 (59) | 90 (98)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
Eczema infantile (Skin and subcutaneous tissue disorders) | 9 (11) | 21 (23)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Ephelides (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Lichen striatus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cataract subcapsular (Eye disorders) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 37 (47) | 60 (71)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (10)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 48 (55) | 93 (108)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (8) | 17 (17)
Rash papular (Skin and subcutaneous tissue disorders) | 8 (8) | 15 (15)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 17 (17) | 40 (40)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Conjunctival hyperaemia (Eye disorders) | 2 (2) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 15 (18)
Thermal burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Transient neonatal pustular melanosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 9 (11) | 21 (25)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria contact (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Circumcision (Surgical and medical procedures) | 1 (1) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 6 (6)
Clamping of blood vessel (Surgical and medical procedures) | 0 (0) | 1 (1)
Infection prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1)
Oral surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Scrotal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin lesion removal (Surgical and medical procedures) | 0 (0) | 1 (2)
Urethral repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Cyanosis (Vascular disorders) | 1 (1) | 3 (3)
Pallor (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 2 (2) | 6 (6)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Hypermetropia (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Lacrimal structural disorder (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Ocular hyperaemia (Eye disorders) | 0 (0) | 4 (4)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0)
Pseudostrabismus (Eye disorders) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 1 (1)
Pupillary disorder (Eye disorders) | 0 (0) | 1 (1)
Strabismus (Eye disorders) | 2 (2) | 3 (3)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 5 (5)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 3 (3) | 6 (6)
Anal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2)
Auriculotemporal syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 38 (42) | 88 (96)
Diarrhoea (Gastrointestinal disorders) | 89 (104) | 171 (196)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epulis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03979313/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT03979313/SAP_001.pdf